CLINICAL TRIAL: NCT04476056
Title: Analysis of Trans-sectoral Nutritional Care of Malnourished Patients With Chronic Pancreatitis Over 6 Months
Brief Title: Malnutrition in Chronic Pancreatitis, Trans-sectoral Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: University of Applied Sciences Neubrandenburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB 069/19
Record Dates: First submitted 2020-06-29; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pancreatitis; Malnutrition; Sarcopenia
MeSH Terms: conditions — Pancreatitis, Chronic; Malnutrition; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic Pancreatitis + Malnutrition (Experimental): Malnourished patients with chronic pancreatitis will receive intensified nutritional therapy for 6 months.
  Interventions: Other: Intensified Nutritional Therapy

INTERVENTIONS:
Other: Intensified Nutritional Therapy — Intensified nutritional therapy will begin in the hospital setting and comprises intake of a commercial oral nutritional supplement (Fortimel Compact 2.4, Nutricia) twice per day as well as personalized dietary counselling. After discharge, supplementation will be continued for at least 28 days and if necessary throughout the entire study duration. Likewise, dietary counselling will be provided throughout the entire study period based on the patient's individual need. Dietary counselling is provided either face-to-face during the follow-up visits or remotely via telephone between visits.

SUMMARY:
Malnutrition and loss of muscle mass are common in patients with chronic pancreatitis. However, there is only limited data on nutritional treatment. In this study, malnourished patients with chronic pancreatitis will receive an intensified nutritional therapy to improve nutritional status. The aim of the study is that malnutrition in patients with chronic pancreatitis can be successfully treated.

DETAILED DESCRIPTION:
Malnutrition and sarcopenia are common complications in chronic pancreatitis leading to increased morbidity and mortality. Therefore nutritional therapy can be considered imperative. However, there is limited evidence on the treatment of malnutrition in patients with chronic pancreatitis. This study aims to investigate the effect of an intensified nutritional therapy on nutritional status in malnourished patients with chronic pancreatitis. By testing feasibility of this intensified therapy valuable recommendations for future treatment of malnutrition in patients with chronic pancreatitis can be derived.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pancreatitis verified by histology or imaging modality (endoscopic ultrasound, computed tomography, magnetic resonance imaging, magnetic resonance cholangiopancreatography)
* Diagnosis of malnutrition

Exclusion Criteria:

* Pregnant or breast feeding
* Implanted defibrillator or pacemaker
* History of pancreatic Cancer
* Any other malignant tumor disease within the last 3 years
* Concomitant liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Malnutrition Status according to ESPEN (European Society for Clinical Nutrition and Metabolism) Criteria | 6 months
  Changes from baseline prevalence of malnutrition according to the European Society for Clinical Nutrition and Metabolism criteria after 6 months

SECONDARY OUTCOMES:
Malnutrition Status according to ESPEN (European Society for Clinical Nutrition and Metabolism) criteria | 28 days, 3 months, 6 months
  Prevalence of malnutrition according to the European Society for Clinical Nutrition and Metabolism criteria
Dropout Rate | 28 days, 3 months, 6 months
  Dropout Rate
Compliance to Oral Nutritional Supplements | 28 days, 3 months, 6 months
  Compliance is assessed by a standardized telephone interview comparing recommended and current intake
Compliance to Dietary Counselling | 28 days, 3 months, 6 months
  Compliance is assessed via standardized telephone interview comparing scheduled and cancelled sessions
Malnutrition according to GLIM (Global Leadership Initiative on Malnutrition) criteria | 28 days, 3 months, 6 months
  Prevalence of malnutrition according to the Global Leadership Initiative on Malnutrition criteria
Sarcopenia according to EWGSOP 2 (European Working Group on Sarcopenia in Older People 2) criteria | 28 days, 3 months, 6 months
  Prevalence of sarcopenia according to the European Working Group on Sarcopenia in Older People 2 criteria
Reduced Body Mass Index | 28 days, 3 months, 6 months
  Changes in prevalence of reduced body mass index (< 18,5 kg/m², < 20 kg/m² if age < 70 yrs, < 22 kg/m² if age ≥ 70 yrs)
Reduced Fat Free Mass Index | 28 days, 3 months, 6 months
  Changes in prevalence of reduced fat free mass index (≤ 15 kg/m² if female, ≤ 17 kg/m² if male)
Reduced Skeletal Muscle Mass Index | 28 days, 3 months, 6 months
  Changes in prevalence of reduced skeletal muscle mass index (≤ 6,42 kg/m² if female, ≤ 8,87 kg/m² if male)
Reduced Gait Speed | 28 days, 3 months, 6 months
  Changes in prevalence of reduced gait speed (< 0,8 m/s)
Reduced Muscle Strength | 28 days, 3 months, 6 months
  Changes in prevalence of reduced muscle strength (< 19,3 kg if female, < 30,3 kg if male)
Body Weight | 28 days, 3 months, 6 months
  Changes in body weight measured in kilograms
Height | 28 days, 3 months, 6 months
  Changes height measured in centimeters
Body Mass Index | 28 days, 3 months, 6 months
  Changes in body mass index measured in kg/m^2 (calculated from the values obtained for body weight and height)
Waist Circumference | 28 days, 3 months, 6 months
  Changes in waist circumference measured in centimeters
Hip Circumference | 28 days, 3 months, 6 months
  Changes in hip circumference measured in centimeters
Waist-to-Hip Ratio | 28 days, 3 months, 6 months
  Changes in waist-to-hip ratio (calculated from the values obtained for waist and hip circumference)
Triceps Skinfold Thickness | 28 days, 3 months, 6 months
  Changes in triceps skinfold thickness measured in millimeters
Upper Arm Circumference | 28 days, 3 months, 6 months
  Changes in upper arm circumference measured in centimeters
Fat Free Mass | 28 days, 3 months, 6 months
  Changes in fat free mass measured by Bioelectrical Impedance Analysis (BIA)
Skeletal Muscle Mass | 28 days, 3 months, 6 months
  Changes in skeletal muscle mass measured by Bioelectrical Impedance Analysis (BIA)
Fat Mass | 28 days, 3 months, 6 months
  Changes in fat mass measured by Bioelectrical Impedance Analysis (BIA)
Total Body Water | 28 days, 3 months, 6 months
  Changes in total body water measured by Bioelectrical Impedance Analysis (BIA)
Extracellular Water | 28 days, 3 months, 6 months
  Changes in extracellular water measured by Bioelectrical Impedance Analysis (BIA)
Phase Angle | 28 days, 3 months, 6 months
  Changes in phase angle measured by Bioelectrical Impedance Analysis (BIA)
Energy Intake | 28 days, 3 months, 6 months
  Changes in energy intake assessed by the German Health Interview and Examination Survey for Adults Food Frequency Questionnaire (DEGS-FFQ)
Protein Intake | 28 days, 3 months, 6 months
  Changes in protein intake assessed by the German Health Interview and Examination Survey for Adults Food Frequency Questionnaire (DEGS-FFQ)
Carbohydrate Intake | 28 days, 3 months, 6 months
  Changes in carbohydrate intake assessed by the German Health Interview and Examination Survey for Adults Food Frequency Questionnaire (DEGS-FFQ)
Fat Intake | 28 days, 3 months, 6 months
  Changes in fat intake assessed by the German Health Interview and Examination Survey for Adults Food Frequency Questionnaire (DEGS-FFQ)
Dietary Fiber Intake | 28 days, 3 months, 6 months
  Changes in dietary fiber intake assessed by the German Health Interview and Examination Survey for Adults Food Frequency Questionnaire (DEGS-FFQ)
Physical Activity | 28 days, 3 months, 6 months
  Changes in metabolic equivalent of task per day and activity level are assessed by employment of the German version of the International Physical Activity Questionnaire (IPAQ) Short Form
Hemoglobin | 28 days, 3 months, 6 months
  Changes in hemoglobin level
Hematocrit | 28 days, 3 months, 6 months
  Changes in hematocrit level
Mean Corpuscular Volume | 28 days, 3 months, 6 months
  Changes in mean corpuscular volume
Mean Corpuscular Hemoglobin Concentration | 28 days, 3 months, 6 months
  Changes in mean corpuscular hemoglobin concentration
Reticulocyte Count | 28 days, 3 months, 6 months
  Changes in reticulocyte count
Sodium | 28 days, 3 months, 6 months
  Changes in plasma concentration of sodium
Potassium | 28 days, 3 months, 6 months
  Changes in plasma concentration of potassium
Calcium | 28 days, 3 months, 6 months
  Changes in plasma concentration of calcium
Magnesium | 28 days, 3 months, 6 months
  Changes in plasma concentration of magnesium
Phosphate | 28 days, 3 months, 6 months
  Changes in plasma concentration of phosphate
Aspartate Transaminase | 28 days, 3 months, 6 months
  Changes in plasma concentration of aspartate transferase
Alanine Aminotransferase | 28 days, 3 months, 6 months
  Changes in plasma concentration of alanine aminotransferase
Gamma-glutamyl Transferase | 28 days, 3 months, 6 months
  Changes in plasma concentration of gamma-glutamyl transferase
Alkaline Phosphatase | 28 days, 3 months, 6 months
  Changes in plasma concentration of alkaline phosphatase
Bilirubin | 28 days, 3 months, 6 months
  Changes in plasma concentration of bilirubin
C-reactive Protein | 28 days, 3 months, 6 months
  Changes in plasma concentration of C-reactive protein
Interleukin-1 Beta | 28 days, 3 months, 6 months
  Changes in serum concentration of interleukin-1 beta
Interleukin-6 | 28 days, 3 months, 6 months
  Changes in plasma concentration of interleukin-6
Tumor Necrosis Factor Alpha | 28 days, 3 months, 6 months
  Changes in serum concentration of tumor necrosis factor alpha
Albumin | 28 days, 3 months, 6 months
  Changes in plasma concentration of albumin
Creatinine | 28 days, 3 months, 6 months
  Changes in plasma concentration of creatinine
Urea | 28 days, 3 months, 6 months
  Changes in plasma concentration of urea
Uric Acid | 28 days, 3 months, 6 months
  Changes in plasma concentration of uric acid
Glucose | 28 days, 3 months, 6 months
  Changes in plasma concentration of glucose
Glycated hemoglobin | 28 days, 3 months, 6 months
  Changes in plasma concentration of glycated hemoglobin
Insulin | 28 days, 3 months, 6 months
  Changes in serum concentration of insulin
Total Cholesterol | 28 days, 3 months, 6 months
  Changes in plasma concentration of total cholesterol
High-density Lipoprotein Cholesterol | 28 days, 3 months, 6 months
  Changes in plasma concentration of high-density lipoprotein cholesterol
Low-density Lipoprotein Cholesterol | 28 days, 3 months, 6 months
  Changes in plasma concentration of high-density lipoprotein cholesterol
Triglycerides | 28 days, 3 months, 6 months
  Changes in plasma concentration of triglycerides
Non-essential Fatty Acids | 28 days, 3 months, 6 months
  Changes in plasma concentration of non-essential fatty acids
Zinc | 28 days, 3 months, 6 months
  Changes in serum concentration of zinc
Iron | 28 days, 3 months, 6 months
  Changes in plasma concentration of iron
Hand Grip Strength | 28 days, 3 months, 6 months
  Changes in maximal hand grip strength
Gait Speed | 28 days, 3 months, 6 months
  Changes in gait speed
Anxiety and Depression | 28 days, 3 months, 6 months
  Changes in anxiety and depression assessed by the German version of the Hospital Anxiety and Depression Scale (HADS-D). For both the anxiety and the depression subscale scores range from 0-21, with higher values indicating a worse outcome.
Fatigue | 28 days, 3 months, 6 months
  Changes in fatigue assessed by the German version of the Fatigue Severity Scale (FSS). Scores range from 1-7, with higher values indicating a better outcome.
Loneliness | 28 days, 3 months, 6 months
  Changes in loneliness assessed by the German Version of the 6-item De Jong Gierveld Loneliness Scale. Scores range from 0-6, with higher values indicating worse outcome.
Intestinal Microbiome | 28 days, 3 months, 6 months
  Changes in the intestinal microbiome
Plasma Metabolome | 28 days, 3 months, 6 months
  Changes in the plasma metabolome
Plasma Transcriptome | 28 days, 3 months, 6 months
  Changes in the plasma transcriptome

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Markus M. Lerch, Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

REFERENCES:
- [Derived] Wiese ML, Frost F, Meyer F, Muller J, Valentini L, Rischmuller K, Lamprecht G, Steveling A, Lerch MM, Aghdassi AA. An intensified trans-sectoral nutritional intervention in malnourished patients with chronic pancreatitis improves diseases prognosis and identifies potential biomarkers of nutritional status. Front Med (Lausanne). 2024 Oct 8;11:1446699. doi: 10.3389/fmed.2024.1446699. eCollection 2024. PMID 39440042